CLINICAL TRIAL: NCT03522194
Title: Influence of Left Ventricular Diastolic Function on Hemodynamic Stability During Anesthesia Induction and on Postoperative Complications
Brief Title: Left Ventricular Diastolic Function During Anesthesia Induction
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV 5436
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Left Ventricular Diastolic Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sevoflurane: Anesthesia maintenance
  Interventions: Drug: Sevoflurane
- Propofol: Anesthesia maintenance
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Sevoflurane — Anesthesia maintenance with Sevoflurane
  Groups: Sevoflurane
Drug: Propofol — Anesthesia maintenance with Propofol
  Groups: Propofol

SUMMARY:
Diastolic dysfunction is an important cause of hemodynamic instability in the perioperative field.Therefore this study aims to investigate the influence of existing diastolic dysfunction or deterioration of diastolic function on hemodynamic stability during induction of anesthesia and postoperative complications. The impact of different anesthetics on diastolic function is investigated.

DETAILED DESCRIPTION:
In this prospective observational study two cohorts of patients with different anesthesia regimes are investigated. Anesthesia is maintained with sevoflurane or propofol. Before induction of anesthesia a transthoracic echocardiography is performed to examine systolic and diastolic function. Immediately after induction, during maintenance and after completion of anesthesia any changes of diastolic function are examined with transthoracic echocardiography. All anesthetic medications, fluids, vasoactive medications and catecholamines are registered.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 60 years scheduled for general anesthesia

Exclusion Criteria:

* Mitral regurgitation or stenosis > I°
* Sp. mitral valve repair or replacement
* Pericardial effusion
* Atrial fibrillation/flutter
* Patients with pacemaker
* BMI > 35 kg/m2

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Norepinephrine | 30 minutes after induction of anesthesia
  Cumulative dose of norepinephrine (adjusted for body weight) during the first 30 minutes after induction of anesthesia

SECONDARY OUTCOMES:
e' | Directly after induction of anesthesia
  Change of the echocardiographic tissue doppler parameter e' after induction of anesthesia
E / e' | Directly after induction of anesthesia
  Change of the echocardiographic index of transmitral flow and tissue doppler after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Katharina Roeher, Dr. med., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Kahl U, Vens M, Pollok F, Menke M, Duckstein C, Gruetzmacher J, Schirren L, Yu Y, Fischer M, Zollner C, Goepfert MS, Roeher K. Do Elderly Patients With Diastolic Dysfunction Require Higher Doses of Norepinephrine During General Anesthesia for Noncardiac Surgeries? A Prospective Observational Study. Anesth Analg. 2021 Feb 1;132(2):420-429. doi: 10.1213/ANE.0000000000005304. PMID 33264119